CLINICAL TRIAL: NCT06934226
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled and Ustekinumab Active Comparator-controlled Study to Evaluate the Efficacy and Safety of JNJ-77242113 for the Treatment of Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Assess Efficacy and Safety of JNJ-77242113 Compared to Placebo and Ustekinumab in Participants With Moderate to Severe Plaque Psoriasis
Acronym: ICONIC-ASCEND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77242113PSO3006; 77242113PSO3006 (Other: Janssen Research & Development, LLC); 2024-515706-77-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1: JNJ 77242113 (Experimental): Participants will receive JNJ-77242113 once daily from Week 0 through Week 104. All participant will receive ustekinumab matching placebo at Week 0, 4 and 16 to maintain the blind.
  Interventions: Drug: JNJ-77242113; Drug: Matching Placebo to Ustekinumab
- Arm 2: Placebo (Placebo Comparator): Participants will receive matching placebo for JNJ-77242113 from Week 0 through Week 16, matching placebo for ustekinumab at Week 0, 4 and 16 and JNJ-77242113 from Week 16 through Week 104.
  Interventions: Drug: JNJ-77242113; Drug: Matching Placebo to JNJ-77242113; Drug: Matching Placebo to Ustekinumab
- Arm 3: Ustekinumab (Active Comparator): Participants will receive Ustekinumab at Week 0, Week 4, and Week 16 followed by JNJ-77242113 once daily from Week 28 through Week 104. Participants will receive both Ustekinumab and placebo for JNJ-77242113 to maintain the blind through Week 28.
  Interventions: Drug: JNJ-77242113; Drug: Matching Placebo to JNJ-77242113; Drug: Ustekinumab

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 will be administered orally.
Drug: Matching Placebo to JNJ-77242113 — Matching placebo will be administered orally.
  Arms: Arm 2: Placebo; Arm 3: Ustekinumab
Drug: Ustekinumab — Ustekinumab will be administered subcutaneously.
  Other Names: STELARA; CNTO 1275
  Arms: Arm 3: Ustekinumab
Drug: Matching Placebo to Ustekinumab — Matching placebo will be administered subcutaneously.
  Arms: Arm 1: JNJ 77242113; Arm 2: Placebo

SUMMARY:
The main purpose of this study is to assess how well JNJ-77242113 works when compared to placebo and ustekinumab in participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis, with or without psoriatic arthritis (PsA), prior to the first administration of study intervention
* Total body surface area (BSA) greater than or equal to (>=)10 percent (%) at screening and baseline
* Total psoriasis area and severity index (PASI) >=12 at screening and baseline
* Total investigator global assessment (IGA) >=3 at screening and baseline
* Candidate for phototherapy or systemic treatment for plaque psoriasis

Exclusion Criteria:

* Nonplaque form of psoriasis (for example [e.g.], erythrodermic, guttate, or pustular)
* Current drug-induced psoriasis (e.g., a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Known allergies, hypersensitivity, or intolerance to JNJ-77242113, ustekinumab, or its excipients
* Major surgical procedure within 8 weeks before screening, or will not have fully recovered from surgical procedure, or has a surgical procedure planned during the time the participant is expected to participate in the study
* Transplanted organ (with exception of a corneal transplant greater than [>] 12 weeks before the first administration of study intervention)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
JNJ-77242113 and Placebo Group: Percentage of Participants with Investigator's Global Assessment (IGA) Score of 0 or 1 and Greater than or Equal to (>=) 2 Grade Improvement from Baseline at Week 16 | Week 16
  IGA score is given based on the investigator's assessment of the participant's plaque psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's plaque psoriasis is assessed as: cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 90 Response at Week 16 | Week 16
  PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In this system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe) and extent of involvement on a scale of 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants achieving at least a 90 percent improvement from baseline in the PASI score.

SECONDARY OUTCOMES:
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving PASI 75 Response at Week 16 | Week 16
  PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In this system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe) and extent of involvement on a scale of 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 75 response represents participants achieving at least a 75 percent improvement from baseline in the PASI score.
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving PASI 100 Response at Week 16 | Week 16
  PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In this system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe) and extent of involvement on a scale of 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 100 response represents participants achieving at least a 100 percent improvement from baseline in the PASI score.
JNJ-77242113 and Placebo Group: Percentage of Participants with IGA Score of 0 at Week 16 | Week 16
  IGA score is given based on the investigator's assessment of the participant's plaque psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's plaque psoriasis is assessed as: cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
JNJ-77242113 and Ustekinumab Group: Percentage of Participants with IGA Score of 0 at Week 28 | Week 28
  IGA score is given based on the investigator's assessment of the participant's plaque psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's plaque psoriasis is assessed as: cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
JNJ-77242113 and Ustekinumab Group: Percentage of Participants Achieving PASI 90 Response at Week 28 | Week 28
  PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In this system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe) and extent of involvement on a scale of 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants achieving at least a 90 percent improvement from baseline in the PASI score.
JNJ-77242113 and Ustekinumab Group: Percentage of Participants Achieving PASI 100 Response at Week 28 | Week 28
  PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In this system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe) and extent of involvement on a scale of 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 100 response represents participants achieving at least a 100 percent improvement from baseline in the PASI score.
JNJ-77242113 and Placebo Group: Percentage of Participants with PSSD Symptom Score of 0 at Week 16 | Week 16
  PSSD includes patient-reported outcome (PRO) questionnaires designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. This PRO includes 11 items in total, with 5 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and 6 items covering participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding). The PSSD itch score will range from 0 to 10. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Percentage of Participants with >= 4 Point Improvement from Baseline in PSSD Itch Score at Week 16 | Week 16
  PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. This PRO includes 11 items in total, with 5 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and 6 items covering participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding). The PSSD itch score will range from 0 to 10. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Number of Participants Reporting Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 108
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. SAE is any untoward medical occurrence that results in: death, is life-threatening, requires in-patient hospitalization/prolongs existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of infectious agent via medicinal product & is medically important.
JNJ-77242113 and Placebo Group: Percentage of Participants with PSSD Sign Score of 0 at Week 16 | Week 16
  PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. This PRO includes 11 items in total, with 6 items covering participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding). A 0 to 10 numerical rating scale for severity is used to rank the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Change from Baseline in Dermatology Life Quality Index (DLQI) Score at Week 16 | Baseline up to Week 16
  DLQI will be utilized in the adult population and is a dermatology specific health related quality of life (HRQoL) instrument designed to assess the impact of the disease on the HRQoL It is a 10-item questionnaire that can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
JNJ-77242113 and Placebo Group: Percentage of Participants with DLQI Score of 0 or 1 at Week 16 | Week 16
  DLQI will be utilized in the adult population and is a dermatology specific HRQoL instrument designed to assess the impact of the disease on the HRQoL It is a 10 item questionnaire that can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
JNJ-77242113 and Placebo Group: Change from Baseline in Body Surface Area (BSA) Score at Week 16 | Baseline up to Week 16
  BSA is a commonly used measure of involvement of skin disease. It is defined as the percentage of surface area of the body involved with the condition being assessed, (that is., plaque psoriasis). The handprint method for assessing BSA will be used, where the surface area of the participant's hand including the palm and all 5 digits is used as a guide to estimate 1% BSA.
JNJ-77242113 and Ustekinumab Group: Percentage of Participants with >= 4 Point Improvement from Baseline in PSSD Itch Score at Week 28 | Week 28
  PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. This PRO includes 11 items in total, with 5 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and 6 items covering participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding). The PSSD itch score will range from 0 to 10. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Ustekinumab Group: Change from Baseline in PSSD Sign Score at Week 28 | Baseline up to Week 28
  PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. This PRO includes 11 items in total, with 5 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and 6 items covering participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding). The PSSD itch score will range from 0 to 10. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Ustekinumab Group: Change from Baseline in PSSD Symptom Score at Week 28 | Baseline up to Week 28
  PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. This PRO includes 11 items in total, with 5 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and 6 items covering participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding). The PSSD itch score will range from 0 to 10. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Ustekinumab Group: Percentage of Participants with PSSD Sign Score of 0 at Week 28 | Week 28
  PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. This PRO includes 11 items in total, with 5 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and 6 items covering participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding). The PSSD itch score will range from 0 to 10. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Ustekinumab Group: Percentage of Participants with PSSD Symptom Score of 0 at Week 28 | Week 28
  PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. This PRO includes 11 items in total, with 5 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and 6 items covering participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding). The PSSD itch score will range from 0 to 10. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Ustekinumab Group: Change from Baseline in DLQI Score at Week 28 | Baseline up to Week 28
  DLQI will be utilized in the adult population and is a dermatology specific HRQoL instrument designed to assess the impact of the disease on the HRQoL It is a 10-item questionnaire that can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
JNJ-77242113 and Ustekinumab Group: Percentage of Participants with DLQI Score of 0 or 1 at Week 28 | Week 28
  DLQI will be utilized in the adult population and is a dermatology specific HRQoL instrument designed to assess the impact of the disease on the HRQoL. It is a 10-item questionnaire that can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
JNJ-77242113 and Ustekinumab Group: Change from Baseline in BSA Score at Week 16 | Baseline up to Week 16
  BSA is a commonly used measure of involvement of skin disease. It is defined as the percentage of surface area of the body involved with the condition being assessed, (ie, plaque psoriasis). The handprint method for assessing BSA will be used, where the surface area of the participant's hand including the palm and all 5 digits is used as a guide to estimate 1% BSA.
JNJ-77242113 and Ustekinumab Group: Percentage of Participants with IGA Score of 0 at Week 16 | Week 16
  IGA score is given based on the investigator's assessment of the participant's plaque psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's plaque psoriasis is assessed as: cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
JNJ-77242113 and Ustekinumab Group: Percentage of Participants Achieving PASI 90 Response at Week 16 | Week 16
  PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In this system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe) and extent of involvement on a scale of 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants achieving at least a 90 percent improvement from baseline in the PASI score.
JNJ-77242113 and Ustekinumab Group: Percentage of Participants Achieving PASI 100 Response at Week 16 | Week 16
  PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In this system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe) and extent of involvement on a scale of 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 100 response represents participants achieving at least a 100 percent improvement from baseline in the PASI score.

CONTACTS AND LOCATIONS:
Locations (160):
- United States (48):
  - Cahaba Research Inc, Birmingham, Alabama
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - T Joseph Raoof Md Inc, Encino, California
  - First OC Dermatology, Fountain Valley, California
  - Dermatologist Medical Group of North County, Inc., Oceanside, California
  - NorCal Clinical Research, Rocklin, California
  - Integrative Skin Science and Research, Sacramento, California
  - MedDerm Associates, San Diego, California
  - Southern California Dermatology, Santa Ana, California
  - Olive View-UCLA Education & Research Institute, Sylmar, California
  - University of Conn Health Center, Farmington, Connecticut
  - Driven Research LLC, Coral Gables, Florida
  - Bioclinical Research Alliance Inc., Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Forcare Clinical Research Inc, Tampa, Florida
  - Hamilton Research LLC, Alpharetta, Georgia
  - Northshore Medical Group, Skokie, Illinois
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - University of Iowa, Iowa City, Iowa
  - Equity Medical, Bowling Green, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - The Derm Institute of West Michigan, Caledonia, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Cleaver Dermatology, Kirksville, Missouri
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Mount Sinai Doctors Dermatology, New York, New York
  - Sadick Research Group, New York, New York
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Optima Research, Boardman, Ohio
  - Apex Dermatology Mayfield Heights, Mayfield Heights, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Clinical Research Philadelphia, Philadelphia, Pennsylvania
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Advanced Research Experts PLLC, Nashville, Tennessee
  - Arlington Research Center, Inc., Arlington, Texas
  - Modern Research Associates PLLC, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Kalo Clinical Research, West Valley City, Utah
  - Frontier Derm Partners CRO, LLC, Mill Creek, Washington
- Argentina (13):
  - Consultora Integral de Salud SRL, Barrio Gral Paz Cba Capital
  - Instituto Medico De Alta Complejidad (IMAC), Buenos Aires
  - Mindout Research, Buenos Aires
  - Instituto de Neumonologia y Dermatologia, Buenos Aires
  - Buenos Aires Skin, CABA
  - Investigaciones Medicas IMOBA SRL, CABA
  - CIPREC, CABA
  - Halitus Instituto Medico S.A. - Dermatologia y Estetica, Caba
  - Mautalen Salud e Investigacion, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Instituto De Especialidades De La Salud SRL, Rosario
  - MR Medicina Reumatologica, San Fernando
  - Instituto de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Australia (8):
  - Monash Medical Centre, Clayton
  - Cornerstone Dermatology, Coorparoo
  - Premier Specialists, Kogarah
  - The Alfred Hospital, Melbourne
  - Royal Melbourne Hospital, Melbourne
  - ISHI dermatology, Mitcham
  - Westmead Hospital, Westmead
  - Veracity Clinical Research, Woolloongabba
- Austria (4):
  - LKH Feldkirch, Feldkirch
  - Kepler Universitatsklinikum GmbH, Linz
  - Universtitatsklinikum St Polten, Sankt Pölten
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Belgium (6):
  - UZ Brussel, Brussels
  - AZ St. Lucas, Ghent
  - Ghent University Hospital, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
  - Dermatologie Maldegem, Maldegem
- Canada (9):
  - Skincare Studio Inc Dermatology Clinical Trials, St. John's, Newfoundland and Labrador
  - CCA Medical Research Corporation, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Lovegrove Dermatology, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - The Centre de recherche Saint-Louis, Québec, Quebec
- Denmark (6):
  - Aalborg Sygehus Syd, Aalborg
  - Aarhus University Hospital, Aarhus
  - Gentofte Hospital, Hellerup
  - Bispebjerg Hospital, København NV
  - Odense University Hospital, Odense
  - Sjællands University hospital, Roskilde
- Germany (14):
  - Klinikum Augsburg, Augsburg
  - Fachklinik Bad Bentheim, Bad Bentheim
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Studienzentrum an der Hase GbR, Bramsche
  - Rosenpark Research GmbH, Darmstadt
  - Medizinische Fakultaet Carl Gustav Carus Technische Universitaet Dresden, Dresden
  - Derma-Study-Center Friedrichshafen GmbH, Friedrichshafen
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Studienzentrum Dr Schwarz Germany, Langenau
  - Dermatologie Mahlow, Mahlow
  - Gemeinschaftspraxis Dres. Quist, Mainz
  - Universitaetsklinikum Muenster, Münster
  - Hautarztpraxis, Witten
- Hungary (11):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Uno Medical Trials Ltd., Budapest
  - Derma-B Kft, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - Synexus Magyarorszag Kft, Gyula
  - Porcika Klinika - Vasarhelyi Sarkanyfu Kft., Hódmezővásárhely
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Bacs-kiskun Megyei Korhaz, Kecskemét
  - Allergo-Derm Bakos Kft., Szolnok
  - Medmare Egeszsegugyi Es Szolgaltato Bt., Veszprém
- Poland (13):
  - Specderm Poznanska sp j, Bialystok
  - Osteo-Medic s.c A. Racewicz, J Supronik, Bialystok
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag
  - Care Clinic Sp z o o, Katowice
  - Specjalistyczny gabinet dermatologiczny Aplikacyjno Badawczy Marek Brzewski Pawel Brzewski Spolka Cywilna, Krakow
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Etyka Osrodek Badan Klinicznych, Olsztyn
  - SOLUMED Centrum Medyczne, Poznan
  - Velocity Skierniewice sp z o o, Skierniewice
  - Magdalena Opadczuk Carpe Diem Centrum Medycyny Estetycznej, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - WroMedica, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (5):
  - Uls Alto Ave - Hosp. Sra. Da Oliveira Guimaraes, Braga
  - Unidade Local De Saude Da Regiao De Leiria Epe, Leiria
  - Uls Sao Jose - Hosp. Sto Antonio Dos Capuchos, Lisbon
  - Hosp. Cuf Descobertas, Lisbon
  - Ulssa Hosp. Santo Antonio, Porto
- Spain (15):
  - Hosp. Gral. Univ. Dr. Balmis, Alicante
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp. Univ. San Cecilio, Granada
  - Grupo Dermatologico Y Estetico Pedro Jaen, Madrid
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. de Manises, Manises
  - Hosp. Clinico Univ. de Santiago, Santiago Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Ntra. Sra. de Valme, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. de La Marina Baixa, Villajoyosa
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
  - Hosp. Univ. Miguel Servet, Zaragoza
- United Kingdom (8):
  - Dudley Group NHS Foundation Trust, Dudley
  - London North West University Healthcare NHS Trust, Harrow
  - The Queen Elizabeth Hospital NHS Foundation Trust, Kings Lynn
  - Guys and St Thomas NHS Foundation Trust, London
  - Royal Berkshire Hospital, Reading
  - Salford Royal Hospital, Salford
  - University Hospital Southampton, Southampton
  - Mid Yorkshire NHS Trust, Wakefield

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency